CLINICAL TRIAL: NCT07039513
Title: EVOLUTION OF D-DIMER AS A MARKER OF BLEEDING RISK ON ECMO
Acronym: ECMOstase2
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9557; 2024-A02754-43 (Other: ANSM)
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: ECMO; Mplementation of a Veno-venous VV or Veno-arterial VA; INTENSIVE CARE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood sampling collection — Collection of an additional of 2.7mL citrate tube of blood for a D-dimer dosage.

SUMMARY:
ECMO (extracorporeal membrane oxygenation) is a life-saving device, used in intensive care to treat severe respiratory or cardiac failure. However, it carries a high risk of serious life-threatening bleeding.

Bleeding complications have been attributed to coagulopathy triggered either by the underlying pathology or by the extracorporeal circuit itself, as well as excessive or inappropriate anticoagulation initiated to prevent thrombotic complications.

The objective of this cohort is to confirm the interest of the evolution of D-dimers as a prognostic marker of serious bleeding events in patients on veno-venous (VV) or veno-arterial (VA) ECMO, and to determine the threshold.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Hospitalized patient in intensive care
* Implementation of a VV or VA ECMO for less than 24 hours
* Patient affiliated to a social protection health insurance scheme
* Non-opposition by the patient or a relative in the event that the patient is not in a state to express his or her non-opposition or inclusion in an emergency procedure in the event that the patient is not in a state to express his or her non-opposition and no relative of the patient can be reached.

Exclusion Criteria:

* Patient on veno-arterial ECMO after cardiac, cardiopulmonary surgery or after placement of a left or biventricular cardiac assist device
* Congenital hemostasis disorder or anatomical abnormality predisposing to bleeding
* Dying patient on the day of inclusion
* Patient under judicial protection
* Patient under guardianship or curatorship
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patient in intensive care with implementation of a VV or VA ECMO for less than 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-27 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
To determine the most discriminating 24-hour D-Dimer increase threshold for predicting a serious bleeding event under ECMO within 24 hours of D-Dimer increase | 1 month
  Difference in D-dimer over 24 hours associated with the occurrence of severe bleeding within 24 hours.

SECONDARY OUTCOMES:
To estimate the predictive performance of the 24-hour increase in D-dimer in the occurrence of a serious bleeding event on ECMO within 24 hours. | 1 month
  Sensitivity (Se)
To estimate the predictive performance of the 24-hour increase in D-dimer in the occurrence of a serious bleeding event on ECMO within 24 hours. | 1 month
  Specificity (Spe)
To estimate the predictive performance of the 24-hour increase in D-dimer in the occurrence of a serious bleeding event on ECMO within 24 hours. | 1 month
  Positive Predictive Value (PPV)
To estimate the predictive performance of the 24-hour increase in D-dimer in the occurrence of a serious bleeding event on ECMO within 24 hours. | 1 month
  Negative Predictive Value (NPV)
To estimate the predictive performance of the 24-hour increase in D-dimer in the occurrence of a serious bleeding event on ECMO within 24 hours. | 1 month
  Positive and Negative Likelihood Ratios of 24-Hour D-Dimer Increase
To estimate the incidence of bleeding and thrombotic complications on ECMO on day 10 | 1 month
  Occurrence of hemorrhagic complications on ECMO on day 10:
  Bleeding events defined by BARC classification, type of bleeding (arterial/venous) and location, transfusions of labile blood products (number/volume/type), other treatments (endoscopy with hemostatic procedure,
To estimate the incidence of bleeding and thrombotic complications on ECMO on day 10 | 1 month
  Occurrence of thrombotic complications on ECMO on day 10:
  Thrombotic and ischemic events: ischemic stroke, limb/extremity ischemia, acute coronary syndrome, ECMO circuit thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive - Réanimation Nouvel Hôpital Civil, Strasbourg, France